CLINICAL TRIAL: NCT06723665
Title: The Exploration of 18F-PSMA-1007 PET/CT Imaging in Prostate Cancer Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Principal Investigator, Chunjing Yu, Director, Affiliated Hospital of Jiangnan University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: LS2024279
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; PET/CT; PSMA-1007; 18F
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 18F-PSMA-1007 (Experimental): Subjects: Patients with suspected or diagnosed prostate cancer, or biochemical recurrence of prostate cancer.
  Over 40 years old (including 40 years old); Informed consent and access to follow-up; To exclude patients who are difficult to receive further diagnosis and treatment because of their serious condition.
  PSMA PET/CT was reviewed 7 days and 3 months after surgery. All patients were followed up once every 3 months to understand the progression and survival of the lesions.
  Interventions: Drug: 18F-PSMA-1007
- 18F-FDG (Active Comparator): The corresponding patients underwent PSMAPET/CT examination within one week before and after routine 18F-FDGPCT/CT imaging (control examination). PCT/CT whole body scan was performed 45min-1h after intravenous injection of the developer, and the image processing was as usual.
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-PSMA-1007 — 18F-PSMA-1007 is administered through a superficial dorsal vein, and the patient is given a dose of about 0.1-0.15mCi/kg
  Arms: 18F-PSMA-1007
Drug: 18F-FDG — 18F-FDG is administered through a superficial dorsal vein, and the patient is given a dose of about 0.1-0.15mCi/kg
  Arms: 18F-FDG

SUMMARY:
micro-PET imaging showed that 18F-PSMA-1007 had similar or even better pharmacokinetics and imaging performance than 18F-DCFPyL. Due to the convenience of synthesis and good imaging performance, 18F-PSMA-1007 is expected to be popularized in clinical practice.The purpose of this study is to evaluate the performance of 18F-PSMA-1007 in diagnosis, differential diagnosis and efficacy monitoring of prostate cancer.

DETAILED DESCRIPTION:
1. Visual analysis of images: describe the location, size, shape and degree of uptake of lesions;
2. Semi-quantitative analysis: the ratio of lesion site uptake to liver uptake was measured by area of interest method (ROI);
3. Comparative analysis: Compared with clinical routine 18F-FDG PET/CT imaging, the advantages of PSMA PET/CT imaging were clarified;
4. Evaluation and analysis of efficacy: before and after treatment, to clarify the early treatment evaluation value of PSMA PET/CT imaging, and compare it with 18F-FDG PET/CT imaging;
5. Prognostic study: Through multi-factor analysis, the relationship between the level of PSMA PET/CT imaging uptake and the prognosis of patients was clarified.

ELIGIBILITY:
Inclusion Criteria:

Prostate cancer is clinically suspected. The patient was diagnosed with prostate cancer by biopsy. Prostate cancer needs to be evaluated after treatment.

Exclusion Criteria:

Patients who did not meet the requirements as assessed by the investigator.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
18F-PSMA-1007 PET/CT and 18F-FDG PCT/CT imaging were compared to determine the advantages of 18F-PSMA-PSMA PET/CT imaging for prostate cancer | 1 day
  For patients receiving 18F-PSMA-1007 PET/CT, 18F-FDG PET/CT imaging was performed, and image visual analysis, semi-quantitative analysis and prognostic study were performed on PET/CT images. To evaluate the diagnosis, staging and prognosis of 18F-PSMA-1007

CONTACTS AND LOCATIONS:
Locations (1):
- Affiated Hospital of Jiangnan University, Wuxi, Jiangsu, China